CLINICAL TRIAL: NCT03877952
Title: A Phase 1 Open-label, Single-dose Study Designed to Assess the Mass Balance Recovery and Metabolite Profile and to Identify Metabolite Structures for [14C]-CORT125281 in Healthy Subjects
Brief Title: Mass Balance Recovery and Metabolite Profile of CORT125281 in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Corcept Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CORT125281-602; 2018-001700-11 (EudraCT Number)
Record Dates: First submitted 2019-03-14; First posted 2019-03-18 (Actual); Last update posted 2019-03-18 (Actual); Status verified 2019-03

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Participants (Experimental): On Day 1, participants will receive a single oral dose of 14C-CORT125281 360 mg (6 X 60 mg capsules) after an overnight fast.
  Interventions: Drug: 14C-CORT125281

INTERVENTIONS:
Drug: 14C-CORT125281 — 14C-CORT125281 360 mg capsule for oral administration containing not more than 2.5 megaBequerel (67 μCi) 14C

SUMMARY:
This study will evaluate the mass balance recovery and metabolite profile, and will identify metabolite structures following a single oral dose of 14C-CORT125281 in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index 18.0 to 30.0 kg/m^2, inclusive
* Provide written informed consent
* Have regular bowel movements (i.e., average stool production of ≥1 and ≤3 stools per day)
* Able to swallow capsules
* Adhere to specified contraception requirements.

Exclusion Criteria:

* Have received any investigational medicine in a clinical research study within the previous 3 months, or CORT125281 at any time
* Have a pregnant partner
* Employees or immediate family members of employees of the study site or Sponsor
* History of abuse of any drug or alcohol, or regularly consume more than 21 units alcohol/week
* Smokers or users of e-cigarettes and nicotine replacement products within the last 6 months
* Occupationally exposed worker, as defined in the Ionising Radiation Regulations 2017; greater than background radiation exposure from other sources exceeding 5 milliSieverts (mSv) in the last 12 months or 10 mSv in the last 5 years
* Clinically significant abnormal results of clinical laboratory safety tests, electrocardiogram, or measurement of heart rate and blood pressure
* History of clinically significant cardiovascular, renal, hepatic, respiratory or gastrointestinal disease, neurological or psychiatric disorder
* History and/or symptoms of adrenal insufficiency or any condition that could be aggravated by glucocorticoid blockade (e.g., an autoimmune disease; allergy requiring treatment)
* Donation or loss of greater than 400 mL of blood within the previous 3 months
* Are taking, or have taken, any prescribed or over-the-counter drug or vitamins/herbal remedies within 1 week (longer restrictions apply for some medicines).

NOTE: Other protocol defined Inclusion/ Exclusion criteria may apply.

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-09-13 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-02 (Actual)

PRIMARY OUTCOMES:
Mass Balance Recovery in Excreta After a Single Oral Dose of 14C-CORT125281 | Until the mass balance criteria for all participants have been met (estimated up to 10 days)

SECONDARY OUTCOMES:
Mass Balance Recovery in Urine After a Single Oral Dose of 14C-CORT125281 | Until the mass balance criteria for all participants have been met (estimated up to 10 days)
Mass Balance Recovery in Feces After a Single Oral Dose of 14C-CORT125281 | Until the mass balance criteria for all participants have been met (estimated up to 10 days)
Plasma Pharmacokinetics (PK) of Total Radioactivity after Oral Dosing: Peak Plasma Concentration (Cmax) | Pre-dose and at pre-specified time points up to Day 8 after dosing
Plasma PK of Total Radioactivity after Oral Dosing: Time from Dosing to Cmax (tmax) | Pre-dose and at pre-specified time points up to Day 8 after dosing
Plasma PK of Total Radioactivity after Oral Dosing: Area Under the Plasma Concentration-time Curve from Zero Time to Time of the Last Measurable Concentration (AUC0-last) | Pre-dose and at pre-specified time points up to Day 8 after dosing
Plasma PK of Total Radioactivity after Oral Dosing: Apparent Elimination Half-life (t1/2) | Pre-dose and at pre-specified time points up to Day 8 after dosing
Plasma PK of Total Radioactivity after Oral Dosing: Mean Residence Time (MRT) | Pre-dose and at pre-specified time points up to Day 8 after dosing
Plasma PK of CORT125281 after Oral Dosing: Cmax | Pre-dose and at pre-specified time points up to Day 8 after dosing
Plasma PK of CORT125281 after Oral Dosing: tmax | Pre-dose and at pre-specified time points up to Day 8 after dosing
Plasma PK of CORT125281 after Oral Dosing: AUC0-last | Pre-dose and at pre-specified time points up to Day 8 after dosing
Plasma PK of CORT125281 after Oral Dosing: t1/2 | Pre-dose and at pre-specified time points up to Day 8 after dosing
Plasma PK of CORT125281 after Oral Dosing: MRT | Pre-dose and at pre-specified time points up to Day 8 after dosing
Distribution of Total Radioactivity into Red Blood Cells after Oral Dosing | Pre-dose and at pre-specified time points up to Day 8 after dosing
Number of CORT125281 Metabolites Accounting for ≥10% of Total Radioactivity Detected in Plasma, Urine, and Feces | Until the mass balance criteria for all participants have been met (estimated up to 10 days)
Percentage of Participants with One or More Adverse Events | Until the mass balance criteria for all participants have been met (estimated up to 10 days)

CONTACTS AND LOCATIONS:
Overall Officials: Sharan Sidhu, MBChB, BAO, MRCS, MFPM, Principal Investigator — Quotient Sciences
Locations (1):
- Quotient Sciences, Ruddington, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No